CLINICAL TRIAL: NCT04620044
Title: Comparison of The Effect of The Kaledo Game and The Nutrition Education Prepared According to Health Belief Model on Weight Loss in Overweight and Obez Children
Brief Title: Kaledo Game and The Nutrition Education Prepared According to Health Belief Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Cahide Çevik, PhD student (researcher), Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AfyonkarahisarUHS; OGU-BAP; 2020-3027 (Other: Osmangazi University)
Record Dates: First submitted 2020-10-22; First posted 2020-11-06 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Childhood Obesity
Keywords: Childhood obesity; Game; Health belief model; Kaledo Game
MeSH Terms: conditions — Pediatric Obesity | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kaledo Game (Experimental): Kaledo game, which is a board game, has been developed to inform children about healthy eating. The aim of this game is to teach children calorie balance through the calorie values of foods. Kaledo game gives children the opportunity to stay motivated and have fun. While children are having fun, they also gain the knowledge necessary for healthy eating behavior change. The game is played with 2-4 people. A game session takes 15-30 minutes Children in the playgroup played 15-30 minutes (1 round) Kaledo game every week for 12 weeks.
  Interventions: Other: Kaledo game
- Education (Experimental): The students in the training group were trained for 20 minutes once a week for 12 weeks. Training subjects were prepared in line with health belief model components.
  The following subjects were included in the training content. What is obesity?Risk factors for obesity, Characteristics of obese individuals, What is a healthy diet?Relationship between unhealthy nutrition and obesity, The consequences of unhealthy diet Health problems caused by obesity, What should be done to prevent and control obesity. How should nutrition be to lose weight? Positive results which show up with weight loss, Barriers to a healthy diet, Ways to reduce and eliminate barriers How to take action to lose weight?, Benefits of weight loss, Success stories in the fight against obesity, How are eating habits changed?, How can we achieve self-efficacy to change eating habits?
  Interventions: Other: Education
- Control (Experimental): There was no intervention in the control group.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Kaledo game — Before starting the study, the height and weight of the children in the play group were measured and their body mass indexes were calculated. Personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale were applied.Then the game sessions were started.Game sessions lasted 12 weeks. After 12 weeks, the height and weight measurements of the students were made and their body mass indexes were calculated. Personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale were applied.
  Arms: Kaledo Game
Other: Education — Before starting the study, the height and weight of the children in the education group were measured and their body mass indexes were calculated. Personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale were applied.Then the education sessions were started.education sessions lasted 12 weeks. After 12 weeks, the height and weight measurements of the students were made and their body mass indexes were calculated. Personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale were applied.
  Arms: Education
Other: No intervention — Body mass indexes were calculated by measuring the height and weight of the students.Personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale were applied.The same measurements and scale applications were repeated after 12 weeks.
  Arms: Control

SUMMARY:
According to the World Health Organization, childhood obesity is the most serious problem of this century. Childhood obesity is an important risk factor for many chronic diseases such as insulin resistance, dyslipidemia, hypertension, diabetes, coronary heart disease.Childhood obesity is a serious public health problem and the public health nurse plays an important role in the prevention of obesity. Especially in schools, positive health behaviors of children should be developed by considering them within the scope of school health. Changing the diet in children will make important contributions to the fight against obesity.In order to change the child's diet, it is necessary to teach the child the correct diet. School is the most appropriate educational environment in which the right nutrition can be learned and permanent behavior change can be established.There is a need for effective methods to teach proper nutrition and to achieve weight loss. The aim of this study was to compare the effect of Kaledo game and nutrition education prepared according to health belief model on weight loss in overweight and obese children. This study is randomized controlled experimental study. There were 2 experiments and a control group in the study. Children in the first experimental group were a play session one day a week, and the second experimental group received 20 minutes of nutrition education once a week. No intervention applied to the control group. Children in all three groups were 0, 3. Month-weight measurements made and personal information form, nutrition self-efficacy scale, nutrition attitude scale and nutrition behavior scale applied.

DETAILED DESCRIPTION:
The population of the study consists of overweight and obese students studying in 5th, 6th and 7th grades of secondary school. However, due to the very large population, 3 secondary schools were selected. It was decided to select a sample from these three secondary schools.The children included in the sample were likely to be in different groups. Also, no intervention would be applied to children in the control group. There could be problems such as children labeling each other. To avoid these problems, the groups are divided into schools. The three schools where the research will be conducted were determined by lot method. The first school formed the Kaledo game group, the second school the nutrition education group, and the third school the control group. BMI was determined by making anthropometric measurements of the children attending these schools. These students were stratified according to their overweight and obese status and gender. According to the power analysis, the minimum sample size for the experimental and control groups was calculated as 57 for each group. In this context, the sample size for each group was planned to consist of 64 people, taking into account incomplete and incorrect data and absenteeism. In this study population, students up to the sample size (n = 64) determined (32 overweight students and 32 obese students) by Power analysis for each school were determined by drawing of lots method. Later, the interventions defined in the groups were initiated.

ELIGIBILITY:
Inclusion Criteria:

* Being studying in the 5th 6th and 7th grade
* BMI percentile value above 85
* Volunteering to participate in research
* Parents' consent

Exclusion Criteria:

* Not being studying in the 5th 6th and 7th grade
* BMI percentile value below 85
* Not being willing to participate in research
* Student's parents not giving consent
* Being on a diet under the control of any specialist or using medication for weight control

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Pre-intervention measurements | first month
  Body Mass Index ( kg/m^2)
Pre-intervention measurements | first month
  nutrition self-efficacy scale to measure nutrition self-efficacy The scale consisting of 15 items has a triple Likert type, single factor structure. Scale items take values in the -1, +1 point range (-1: not sure, 0: somewhat sure, +1: very sure). The total score is between -15 and +15. The higher the total score obtained from the scale indicates the high self-efficacy value.
Pre-intervention measurements | first month
  nutrition attitude scale to measure nutrition attitude Scale items take values between 1-4 points (1- strongly disagree, 2- disagree, 3-agree, 4- strongly agree). Its total score is between 4-16. A high total score from the scale indicates a positive attitude.
Pre-intervention measurements | first month
  nutrition behavior scale to measure nutrition behavior Scale items take -1 value for unhealthy food and +1 value for healthy food, total score is between -14, +14. The high total score obtained from the scale indicates the healthy eating habits.

SECONDARY OUTCOMES:
Post-intervention measurements | 3rd month
  Body Mass Index ( kg/m^2)
Post-intervention measurements | 3rd month
  nutrition self-efficacy scale to measure nutrition self-efficacy The scale consisting of 15 items has a triple Likert type, single factor structure. Scale items take values in the -1, +1 point range (-1: not sure, 0: somewhat sure, +1: very sure). The total score is between -15 and +15. The higher the total score obtained from the scale indicates the high self-efficacy value.
Post-intervention measurements | 3rd month
  nutrition attitude scale to measure nutrition attitude Scale items take values between 1-4 points (1- strongly disagree, 2- disagree, 3-agree, 4- strongly agree). Its total score is between 4-16. A high total score from the scale indicates a positive attitude.
Post-intervention measurements | 3rd month
  nutrition behavior scale to measure nutrition behavior Scale items take -1 value for unhealthy food and +1 value for healthy food, total score is between -14, +14. The high total score obtained from the scale indicates the healthy eating habits.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem ÖRSAL, PhD, Study Director — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen M, Uzuner A, Akman M, Bahadir AT, Borekci NO, Viggiano E. Examination of a board game approach to children's involvement in family-based weight management vs. traditional family-based behavioral counseling in primary care. Eur J Pediatr. 2018 Aug;177(8):1231-1238. doi: 10.1007/s00431-018-3177-z. Epub 2018 May 29. PMID 29845514
- [Background] Viggiano A, Viggiano E, Di Costanzo A, Viggiano A, Andreozzi E, Romano V, Rianna I, Vicidomini C, Gargano G, Incarnato L, Fevola C, Volta P, Tolomeo C, Scianni G, Santangelo C, Battista R, Monda M, Viggiano A, De Luca B, Amaro S. Kaledo, a board game for nutrition education of children and adolescents at school: cluster randomized controlled trial of healthy lifestyle promotion. Eur J Pediatr. 2015 Feb;174(2):217-28. doi: 10.1007/s00431-014-2381-8. Epub 2014 Jul 22. PMID 25048788
- [Background] Haney MO, Erdogan S. Factors related to dietary habits and body mass index among Turkish school children: a Cox's interaction model-based study. J Adv Nurs. 2013 Jun;69(6):1346-56. doi: 10.1111/j.1365-2648.2012.06126.x. Epub 2012 Aug 22. PMID 22909283
- [Background] Amaro S, Viggiano A, Di Costanzo A, Madeo I, Viggiano A, Baccari ME, Marchitelli E, Raia M, Viggiano E, Deepak S, Monda M, De Luca B. Kaledo, a new educational board-game, gives nutritional rudiments and encourages healthy eating in children: a pilot cluster randomized trial. Eur J Pediatr. 2006 Sep;165(9):630-5. doi: 10.1007/s00431-006-0153-9. Epub 2006 May 30. PMID 16733670